CLINICAL TRIAL: NCT00537433
Title: An RCT to Reduce Liquid Medication Dosing Errors and Improve Adherence in Caregivers of Young Children Through a Pictogram-Based Intervention
Brief Title: Improving Parental Understanding of Medication Instructions Through a Pictogram-Based Intervention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB06-168
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2007-09

CONDITIONS: Medication Errors
Keywords: Medication errors; Patient nonadherence; Literacy; Communication
MeSH Terms: conditions — Patient Compliance; Literacy; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard counseling (No Intervention): Families in the control group receive standard care, including routine counseling regarding medications prescribed from their physician and post-visit counseling by the pediatric nursing staff. Dosing instruments are given at the discretion of the physician or nurse.
- Pictogram (Experimental): Parents randomized to the pictogram-based intervention group receive medication counseling utilizing the pictogram-based medication instruction sheets. These sheets help to facilitate medication counseling, including teaching about dosage and adherence.
  Interventions: Other: Pictogram

INTERVENTIONS:
Other: Pictogram — The plain language, pictogram-based medication instruction sheets (available in English and Spanish) utilize pictograms to convey information about the medication name, indication, dose, dose frequency, and length of treatment, along with information about preparation and storage. The sheets also include a medication log for parents to keep track of when they administer the medication.
  Research staff reference the sheets as they demonstrate dosing with a standardized dosing instrument; teachback is performed to reinforce concepts. For medications in which a standardized dosing instrument was not included at dispensing, a standardized oral dosing syringe is provided for the caregiver to use at home. After counseling, the caregiver is given the instruction sheet to take home.
  Arms: Pictogram

SUMMARY:
Liquid medication administration errors are common, and place children at risk for adverse events. Caregivers with low socioeconomic status (SES), low education and poor health literacy skills are at increased risk for errors. In this study, we seek to assess whether at-risk parents who received a plain language, pictogram-based intervention would have reduced medication dosing errors and improved medication adherence.

DETAILED DESCRIPTION:
Evidence suggests that errors by parents and caregivers in administering medications to their children are frequent. These errors, which include inaccurate dosing as well as nonadherence to medication regimens, place children at risk for morbidity and mortality. Misdosing is prevalent, with 50% or more of pediatric caregivers either measuring an incorrect dose or reporting a dose of liquid medication given outside the recommended range. Of further concern are reports of an overall poor adherence rate of 50% for pediatric medications, with implications for treatment failure and drug resistance.

Few studies have examined strategies for decreasing medication administration errors in pediatric patients. Pictograms represent a promising approach in which simple diagrams are used to improve understanding of concepts. Pictorial-enhanced written materials have been shown to improve comprehension and adherence with medical directions, particularly for patients with low literacy.

We developed a pictogram-based intervention to decrease dosing errors and improve adherence. In this study, we sought to assess whether this intervention would reduce medication dosing errors and improve adherence in a pediatric emergency room serving at-risk families.

ELIGIBILITY:
Inclusion Criteria:

* child 30 days through 8 years old
* child prescribed a liquid medication (short course (<14 days) daily dose medication or as needed (prn) medication)

Exclusion Criteria:

* caregiver accompanying child to visit not primarily responsible for administering medication to the child
* caregiver not fluent in English or Spanish
* child requiring immediate medical attention
* child who typically takes medications in tablet form
* child having a visit involving a psychiatric problem or child protection issue

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2006-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Medication Dosing Accuracy (observed and reported); Medication Adherence (reported) | Assessments by phone or in-person, planned at 3-5 days for prn medications, and within 1 day of last dose of prescribed treatment time for daily dose medications.

SECONDARY OUTCOMES:
Medication Knowledge and Related Medication Practices (dose frequency, preparation, storage, dosing instrument use) | Assessments by phone or in-person, planned at 3-5 days for prn medications, and within 1 day of last dose of prescribed treatment time for daily dose medications.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang (Shonna) Yin, MD, MS, Principal Investigator — NYU School of Medicine Department of Pediatrics; Alan L Mendelsohn, MD, Principal Investigator — NYU School of Medicine Department of Pediatrics; Benard P Dreyer, MD, Principal Investigator — NYU School of Medicine Department of Pediatrics
Locations (1):
- NYU School of Medicine Department of Pediatrics, New York, New York, United States

REFERENCES:
- [Derived] Yin HS, Dreyer BP, van Schaick L, Foltin GL, Dinglas C, Mendelsohn AL. Randomized controlled trial of a pictogram-based intervention to reduce liquid medication dosing errors and improve adherence among caregivers of young children. Arch Pediatr Adolesc Med. 2008 Sep;162(9):814-22. doi: 10.1001/archpedi.162.9.814. PMID 18762597